CLINICAL TRIAL: NCT02470377
Title: Transcranial Magnetic Stimulation for Mal de Debarquement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Principal Investigator, Yoon-Hee Cha, Yoon-Hee Cha, MD, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-003-01
Record Dates: First submitted 2015-06-09; First posted 2015-06-12 (Estimated); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Mal de Debarquement Syndrome
Keywords: MdDS; TMS; fMRI; EEG
MeSH Terms: conditions — Mal de debarquement | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This was an N-of-1 pilot study in which all participants received one session of each of 3 targets and chose which of the 3 led to the most acute reduction in intensity of rocking. The participants were treated with the target that they chose and then completed post stimulation diaries.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Target 1: Occipital Cortex (Experimental): After determination of the motor threshold, the TMS coil will be positioned over the midline occipital cortex using MRI guidance and a frameless stereotaxy system. A train of stimulation pulses in continuous theta burst mode will be delivered.
  Interventions: Device: Transcranial Magnetic Stimulation
- Target 2: Cerebellar Vermis (Experimental): After determination of the motor threshold, the TMS coil will be positioned over the midline cerebellar vermis using MRI guidance and a frameless stereotaxy system. A train of stimulation pulses in continuous theta burst mode will be delivered.
  Interventions: Device: Transcranial Magnetic Stimulation
- Target 3: Cerebellar Hemisphere (Active Comparator): After determination of the motor threshold, the TMS coil will be positioned over the lateral cerebellar hemisphere using MRI guidance and a frameless stereotaxy system. A train of stimulation pulses in continuous theta burst mode will be delivered.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.

SUMMARY:
The goal of this study is to determine whether external neuromodulation using repetitive transcranial magnetic stimulation (rTMS) can reduce the perception of self-motion that is experienced by individuals with mal de debarquement syndrome (MdDS). Mal de debarquement is translated as the "sickness of disembarkment," and refers to the chronic feeling of rocking dizziness that occurs after exposure to passive motion. Treatment for MdDS is limited and morbidity is high. The goal of the study is to determine whether rTMS can suppress the rocking dizziness of MdDS.

DETAILED DESCRIPTION:
Participants will maintain web-based diaries of their symptoms for two weeks prior to treatment with rTMS. Up to 20 treatments with rTMS with either anatomically or functionally determined targets will be administered. Post treatment diaries will continue for up to 12 weeks after rTMS administration.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 years old
2. Willing and capable of interacting with the informed consent process
3. Primary disorder being a persistent rocking dizziness triggered by passive motion such as from water, land, or air travel and with no other central nervous system or peripheral vestibular disorder determined after appropriate evaluation.

Exclusion criteria:

1. Subjects who cannot comply with study conditions.
2. Active psychiatric condition such as mania or psychosis
3. Unstable medical condition
4. Implanted metal anywhere in the body (infusion pumps, pacemakers, metal or shrapnel in the body, deep brain stimulators, aneurysm clips, metal prostheses, joints, rods or plates). Dental fillings are acceptable.
5. Personal history of seizures or a first-degree relative with epilepsy
6. Medications known to lower seizure threshold such as: typical (high-potency) neuroleptics and tricyclic antidepressants: Subjects who take one or a combination of the following drugs will be excluded: imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine. clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine (including MDMA, ecstasy), phencyclidine (PCP, angel's dust), ketamine, gamma-hydroxybutyrate (GHB), theophylline, haloperidol, fluphenazine, bupropion.
7. Pregnancy or planning to become pregnant during study enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Hee Cha, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized data may be shared with other researchers when there is sufficient recruitment to assure that no individual may be identified based on demographic or clinical characteristics.

REFERENCES:
- [Result] Cha YH, Ding L, Yuan H. Neuroimaging Markers of Mal de Debarquement Syndrome. Front Neurol. 2021 Mar 4;12:636224. doi: 10.3389/fneur.2021.636224. eCollection 2021. PMID 33746890
- [Result] Cha YH, Gleghorn D, Doudican B. Occipital and Cerebellar Theta Burst Stimulation for Mal De Debarquement Syndrome. Otol Neurotol. 2019 Oct;40(9):e928-e937. doi: 10.1097/MAO.0000000000002341. PMID 31436631
- [Result] Chen Y, Cha YH, Gleghorn D, Doudican BC, Shou G, Ding L, Yuan H. Brain network effects by continuous theta burst stimulation in mal de debarquement syndrome: simultaneous EEG and fMRI study. J Neural Eng. 2021 Nov 30;18(6):10.1088/1741-2552/ac314b. doi: 10.1088/1741-2552/ac314b. PMID 34670201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: August 15 to July 2017
Pre-assignment Details: All enrolled participants were included. This was an N-of-1 study so all participants received one session each of each target. Two participants were excluded prior to enrollment (one due to medical illness before she selected a target, one due to side effects from all targets and not being treated on the protocol).
Groups:
- Occipital Transcranial Magnetic Stimulation: After determination of the motor threshold, the TMS coil will be positioned at predetermined locations over the brain using MRI guidance and a frameless stereotaxy system. A train of continuous theta burst mode will be delivered over the midline occipital cortex with MRI guided neuronavigation.
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
- Cerebellar Vermis Transcranial Magnetic Stimulation: An active comparator not at the target of interest will be used for the study. A train of continuous theta burst mode will be delivered over the midline cerebellar vermis with MRI guided neuronavigation.
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
- Cerebellar Hemisphere Control Transcranial Magnetic Stimulation: An active comparator not at the target of interest will be used for the study. A train of continuous theta burst mode will be delivered over the cerebellar hemisphere with MRI guided neuronavigation.
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
Period: Overall Study
Arm/Group | Occipital Transcranial Magnetic Stimulation | Cerebellar Vermis Transcranial Magnetic Stimulation | Cerebellar Hemisphere Control Transcranial Magnetic Stimulation
Started | 10 | 9 | 5
Completed | 10 | 9 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was an N-of-1 study. The numbers in each treatment category reflect the target that the participant chose after receiving one session each of the three targets given in randomized order.
Groups:
- Target 1: Occipital Cortex: After determination of the motor threshold, the TMS coil will be positioned at predetermined locations over the brain using MRI guidance and a frameless stereotaxy system. A train of continuous theta burst mode will be delivered at the midline occipital cortex, with the brain locations determined by MRI and real-time neuronavigation.
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
- Target 2: Cerebellar Vermis: An active comparator not at the target of interest will be used for the study. A train of continuous theta burst mode will be delivered at the midline cerebellar vermis, with the brain locations determined by MRI and real-time neuronavigation.
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
- Target 3: Cerebellar Hemisphere: An active comparator not at the target of interest will be used for the study. A train of continuous theta burst mode will be delivered at the cerebellar hemisphere with the brain locations determined by MRI and real-time neuronavigation.
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
- Total: Total of all reporting groups
Arm/Group | Target 1: Occipital Cortex | Target 2: Cerebellar Vermis | Target 3: Cerebellar Hemisphere | Total
Number analyzed (Participants) | 10 | 9 | 5 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (11.1) | 53.6 (11.5) | 42.6 (14.0) | 51.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 5 | 24
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 9 | 5 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Dizziness Handicap Inventory Total [Mean (Standard Deviation); unit: units on a scale] — The Dizziness Handicap Inventory is a widely used measure of subjective dizziness in which 25 questions of dizziness inducing events are rated on a scale of 0-2-4. The maximum number of points is 100 points which are divided into the following levels: 16-34 Points (mild handicap), 36-52 Points (moderate handicap), 54+ Points (severe handicap).
  Results reported are the differences immediately and at 6 weeks post-stimulation from the mean of the baseline 4 weeks of pre-stimulation scores.
  units on a scale | 46.2 (13.7) | 51.1 (13.0) | 51.6 (12.6) | 49.2 (12.9)
Mal de Debarquement Balance Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The MdDS Balance Rating Scale is a 10-point scale inquiring about the severity of rocking vertigo in which 1 means no rocking and 10 is so severe that standing is not possible. A level of 6 indicates that gait is impaired due to the severity of rocking.
  Results reported are the differences immediately and at 6 weeks post-stimulation from the mean of the baseline 4 weeks of pre-stimulation scores.
  units on a scale | 4.6 (1.3) | 5.2 (0.8) | 4.4 (1.5) | 4.8 (1.2)
Hospital Anxiety and Depression Scale-Anxiety [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale is a widely used scale that inquires about anxiety and depression symptoms with 14 questions divided into 7 questions about anxiety and 7 questions about depression. Each item is rated from 0-3 per item yielding a maximum of 21 points per item. Each subscale is rated as follows: 0-7 (Normal), 8-10 (Borderline), 11-21 (Abnormal).
  Results reported are the differences immediately and at 6 weeks post-stimulation from the mean of the baseline 4 weeks of pre-stimulation scores.
  units on a scale | 6.2 (2.6) | 6.3 (3.8) | 9.4 (3.2) | 6.9 (3.3)
Hospital Anxiety and Depression Scale-Depression [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale is a widely used scale that inquires about anxiety and depression symptoms with 14 questions divided into 7 questions about anxiety and 7 questions about depression. Each item is rated from 0-3 per item yielding a maximum of 21 points per item. Each subscale is rated as follows: 0-7 (Normal), 8-10 (Borderline), 11-21 (Abnormal).
  Results reported are the differences immediately and at 6 weeks post-stimulation from the mean of the baseline 4 weeks of pre-stimulation scores.
  units on a scale | 7.0 (3.4) | 8.0 (3.2) | 9.6 (3.8) | 7.9 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Dizziness Handicap Inventory
Description: The Dizziness Handicap Inventory is a widely used measure of subjective dizziness in which 25 questions of dizziness inducing events are rated on a scale of 0-2-4. The maximum number of points is 100 points which are divided into the following levels: 16-34 Points (mild handicap), 36-52 Points (moderate handicap), 54+ Points (severe handicap).
Time Frame: 10 weeks (4 pre stimulation + 6 post stimulation)
Population: The median of the 4 pre-stimulation scores was used as the baseline. The difference between this number and the post-stimulation scores were calculated for each participant. The mean and standard deviation for the change in scores from the median of the baseline scores is presented for each treatment group for scores reported immediately after TMS and 6 weeks post TMS.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Occipital Transcranial Magnetic Stimulation: After determination of the motor threshold, the TMS coil will be positioned at predetermined locations over the brain using MRI guidance and a frameless stereotaxy system. A train of stimulation pulses (repetitive TMS) at 1Hz up to 10Hz or in theta burst mode will be delivered at one or more locations over the head, depending on the brain location under study (brain locations determined by MRI data).
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
- Vermis Transcranial Magnetic Stimulation; Cerebellar Hemisphere Control Transcranial Magnetic Stimulation: An active comparator not at the target of interest will be used for the study.
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
Arm/Group | Occipital Transcranial Magnetic Stimulation | Vermis Transcranial Magnetic Stimulation | Cerebellar Hemisphere Control Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 9 | 5
score on a scale
  Immediate change | -17.5 (10.3) | -3.7 (10.6) | -8.4 (14.4)
  6 week change | -10.1 (18.0) | -9.7 (12.2) | -4.0 (9.0)
Statistical Analysis 1: Comparison: Occipital Transcranial Magnetic Stimulation vs Vermis Transcranial Magnetic Stimulation vs Cerebellar Hemisphere Control Transcranial Magnetic Stimulation; This was an N-of-1 pilot study in which all participants received one session of each of 3 targets and chose which of the 3 led to the most acute reduction in intensity of rocking. The participants were treated with the target that they chose and then completed post stimulation diaries; Test type: Superiority — The hypothesis was that either Target 1 (Occipital) or Target 2 (Vermis) would be more effective than the control target (Cerebellar hemisphere) but that there may be baseline differences in participants who chose Target 1 vs Target 2; p = 0.0439, ANOVA — Only p-values <0.05 were considered significant; One way ANOVA, immediate DHI changes used for calculation

2. Secondary Outcome: Mal de Debarquement Balance Rating Scale
Description: The MdDS Balance Rating Scale is a 10-point scale inquiring about the severity of rocking vertigo in which 1 means no rocking and 10 is so severe that standing is not possible. A level of 6 indicates that gait is impaired due to the severity of rocking.
Time Frame: 10 weeks (4 pre stimulation + 6 post stimulation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Occipital Transcranial Magnetic Stimulation | Vermis Transcranial Magnetic Stimulation | Cerebellar Hemisphere Control Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 9 | 5
score on a scale
  Immediate change | -1.8 (1.3) | -1.3 (0.9) | -0.1 (0.5)
  6 week change | -1.1 (1.7) | -1.3 (1.6) | -0.1 (0.5)
Statistical Analysis 1: Comparison: Occipital Transcranial Magnetic Stimulation vs Vermis Transcranial Magnetic Stimulation vs Cerebellar Hemisphere Control Transcranial Magnetic Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0316, ANOVA; One way ANOVA, immediate MBRS changes used for calculation

3. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: The Hospital Anxiety and Depression Scale is a widely used scale that inquires about anxiety and depression symptoms with 14 questions divided into 7 questions about anxiety and 7 questions about depression. Each item is rated from 0-3 per item yielding a maximum of 21 points per item. Each subscale is rated as follows: 0-7 (Normal), 8-10 (Borderline), 11-21 (Abnormal).
Time Frame: 10 weeks (4 pre stimulation + 6 post stimulation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Occipital Transcranial Magnetic Stimulation | Vermis Transcranial Magnetic Stimulation | Cerebellar Hemisphere Control Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 9 | 5
score on a scale
  Immediate change-Anxiety | -2.5 (2.4) | 0.8 (5.3) | -0.2 (2.6)
  6 week change-Anxiety | -2.2 (2.4) | -1.6 (3.5) | -0.4 (1.9)
  Immediate change-Depression | -2.4 (2.5) | -0.4 (4.9) | 1.4 (2.5)
  6 week change-Depression | -1.7 (4.3) | -1.4 (3.7) | 0.4 (1.0)
Statistical Analysis 1: Comparison: Occipital Transcranial Magnetic Stimulation vs Vermis Transcranial Magnetic Stimulation vs Cerebellar Hemisphere Control Transcranial Magnetic Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1754, ANOVA; One way ANOVA, immediate HADS changes used for calculation

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Target 1 Transcranial Magnetic Stimulation: After determination of the motor threshold, the TMS coil will be positioned at predetermined locations over the brain using MRI guidance and a frameless stereotaxy system. A train of stimulation pulses (repetitive TMS) at 1Hz up to 10Hz or in theta burst mode will be delivered at one or more locations over the head, depending on the brain location under study (brain locations determined by MRI data).
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
- Target 2 Transcranial Magnetic Stimulation; Target 3 Control Site Transcranial Magnetic Stimulation: An active comparator not at the target of interest will be used for the study.
  Transcranial Magnetic Stimulation: A form of external neuromodulation using pulsatile magnetic fields on the surface of the head.
Arm/Group | Target 1 Transcranial Magnetic Stimulation | Target 2 Transcranial Magnetic Stimulation | Target 3 Control Site Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT02470377/Prot_SAP_000.pdf